CLINICAL TRIAL: NCT05406388
Title: Ultrasound-guided Bilateral Erector Spinalis Plane Block on Postoperative Pain Management in Liver Transplantation Donors
Brief Title: Erector Spinae Plane Block in Liver Transplantation Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tumay Uludag Yanaral, Assistant professor, MD, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEDIPOLU-973
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: There are two model for this study. The first group is erector spinae plane block group. The second one is control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Erector Spinae Plane Block for Postoperative Analgesia
  Interventions: Procedure: Erector Spinae Plane Block
- Control group (Active Comparator): No regional anesthesia technique will be applied to the control group.
  Interventions: Procedure: Intravenous fentanyl patient control device

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Intravenous fentanyl patient control device 48-hour fentanyl consumption will be recorded.
  Arms: Erector Spinae Plane Block
Procedure: Intravenous fentanyl patient control device — Intravenous fentanyl patient control device 48-hour fentanyl consumption will be recorded.
  Arms: Control group

SUMMARY:
Living donor liver transplantation has become a common treatment option for patients with end-stage liver disease. Donor hepatectomy is associated with significant postoperative pain due to inverted L-shaped incision. Therefore adequate analgesia is important for recovery.

Erector Spinae Plane Block (ESPB) is a safe anesthesia technique used to provide postoperative analgesia. This study aimed to compare the novel ultrasound-guided ESPB technique with controls in terms of postoperative opioid consumption and postoperative pain control on donor patients.

ELIGIBILITY:
Inclusion Criteria:

* Donor patients scheduled for elective hepatectomy in liver transplantation surgery
* ASA I-II
* Patients who are aged between 18-65

Exclusion Criteria:

* Patients who do not accept the procedure
* Skin infection at the site of Erector Spina Plan Block area
* Coagulation disorder or using anticoagulant drugs
* Known local anesthetics and opioid allergy
* Severe pulmonary and/or cardiovascular problems
* Substance addiction or known psychiatric or mental problems
* Chronic painkiller usage
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 0, 2, 4, 6, 12, 24, 36 and 48 hours
  The amount of fentanyl required by the patient and given by the device will be recorded for the first 48 hours.

SECONDARY OUTCOMES:
Visual Analog Scale | Change from baseline pain scores at postoperative 0, 2, 4, 6, 12, 24, 36 and 48 hours
  Pain of patients will be evaluated and recorded according to the Visual Analog Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tumay Uludag Yanaral, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewe G, Steyaert A, De Kock M, Lois F, Reding R, Forget P. Pain management in living related adult donor hepatectomy: feasibility of an evidence-based protocol in 100 consecutive donors. BMC Res Notes. 2018 Nov 26;11(1):834. doi: 10.1186/s13104-018-3941-1. PMID 30477577
- [Background] Chhibber A, Dziak J, Kolano J, Norton JR, Lustik S. Anesthesia care for adult live donor hepatectomy: our experiences with 100 cases. Liver Transpl. 2007 Apr;13(4):537-42. doi: 10.1002/lt.21074. PMID 17394151
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] El-Boghdadly K, Pawa A. The erector spinae plane block: plane and simple. Anaesthesia. 2017 Apr;72(4):434-438. doi: 10.1111/anae.13830. Epub 2017 Feb 11. No abstract available. PMID 28188611
- [Background] Hacibeyoglu G, Topal A, Arican S, Kilicaslan A, Tekin A, Uzun ST. USG guided bilateral erector spinae plane block is an effective and safe postoperative analgesia method for living donor liver transplantation. J Clin Anesth. 2018 Sep;49:36-37. doi: 10.1016/j.jclinane.2018.06.003. Epub 2018 Jun 5. No abstract available. PMID 29883965